CLINICAL TRIAL: NCT00979693
Title: Psilocybin-assisted Psychotherapy in the Management of Anxiety Associated With Stage IV Melanoma.
Brief Title: Psilocybin-Assisted Psychotherapy for Anxiety in People With Stage IV Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was suspended because the PI was unable to get permission from his department to submit the protocol to the local IRB?"
Sponsor: Multidisciplinary Association for Psychedelic Studies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCA1
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Anxiety; Stage IV Melanoma
Keywords: anxiety; stage IV melanoma; depression; spirituality; pain
MeSH Terms: conditions — Anxiety Disorders; Melanoma; Depression; Pain | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Dose (Experimental): Participant will receive 25 mg psilocybin during two day-long sessions of psychotherapy in combination with psilocybin, with each session scheduled seven to 14 days apart.
  Interventions: Drug: psilocybin
- Active Placebo (Active Comparator): The participant will receive 4 mg psilocybin during two day-long sessions of psychotherapy in combination with psilocybin, with sessions scheduled seven to 14 days apart.
  Interventions: Drug: psilocybin

INTERVENTIONS:
Drug: psilocybin — 25 mg psilocybin administered orally once during each of the two day-long psychotherapy sessions.
  Arms: Full Dose
Drug: psilocybin — 4 mg psilocybin orally administered once during each of two day-long psychotherapy session
  Arms: Active Placebo

SUMMARY:
This study is to find out about whether two sessions of psilocybin-assisted psychotherapy are safe and will help people who are anxious as a result of having stage IV melanoma and will involve two sessions of psychotherapy combined with either 4 or 25 mg psilocybin. The study will measure anxiety, depression, quality of life and spirituality before and after psilocybin-assisted psychotherapy, natural killer cells (a type of immune cell) will be counted from blood samples taken the day after psilocybin-assisted psychotherapy, and people will keep daily diaries reporting on how anxious they feel for each day in the study.

DETAILED DESCRIPTION:
Melanoma is a cancer arising from pigment-producing cells, or melanocytes. These cells are chiefly located in the skin, but they can also be found in other parts of the body, including eyes, ears and GI tract. A diagnosis of stage IV melanoma can create great stress and anxiety for an individual and his or her caregivers. Psilocybin (4-phosphoryloxy- N,N-dimethyl-tryptamine) is a psychedelic (hallucinogenic) compound found in certain species of mushrooms that can produce spiritual or mystical experiences and that has been used in psychotherapy prior to being made illegal. This study will be a randomized, active-placebo controlled pilot study of the safety and efficacy of psilocybin-assisted psychotherapy as a means of managing anxiety in association with stage IV melanoma. This study will examine whether two sessions of psilocybin-assisted psychotherapy scheduled seen to 14 days apart will reduce anxiety, improve quality of life and be safe in people with stage IV melanoma.

Subjects in this study will have a 66% chance of receiving the full dose of 25 mg psilocybin and a 33% of receiving 4 mg psilocybin. The first dose is expected to change how people feel, think and see the world, while the lower dose is expected to have only slight effects. Each subject will receive these conditions at random, as if by coin-toss. The researchers, including the therapists, and the subject will not know whether they are assigned to get 25 or 4 mg psilocybin.

The entire study can last up to three and a half months (14 weeks) but the main part of the study lasts six weeks. After the researchers determine that a person with stage IV melanoma and anxiety can be in the study, there will be two introductory psychotherapy sessions with the therapist-investigators. They will prepare the participant for psilocybin-assisted psychotherapy. The subject will have a day-long psilocybin-assisted psychotherapy session after introductory sessions, and he or she will remain overnight at the clinic. There will be a psychotherapy follow-up scheduled the day after each psilocybin-assisted session to help people work with the psilocybin-assisted psychotherapy, and there will be a psychotherapy session in between the first and second psilocybin-assisted psychotherapy sessions. Two weeks after the second psilocybin-assisted psychotherapy session, subjects will return for another follow-up visit. The subjects will answer questions or fill out questionnaires about anxiety, depression, quality of life, spirituality and sense of self at the start of the study, two weeks after the second psilocybin-assisted session and at least once during the study. Subjects will have blood draws to assess liver function before each psilocybin-assisted session and they will have a blood draw to assess natural killer (NK) cells the day after each psilocybin-assisted session. On the day after each psilocybin-assisted session, subjects will also complete a questionnaire about their experiences during the psilocybin-assisted session.

Two weeks after the second experimental psilocybin-assisted session, subjects will learn if they got the full or active placebo dose of psilocybin. Any of the three subjects who receive the active placebo dose can take part in an "open-label" study phase that will last another six weeks. The open-label phase will be nearly identical to those used in the first study phase except that there will be one, and not two, introductory psychotherapy sessions, and the subject and therapists will know that the subject will be receiving 25 mg psilocybin. People who got the full dose of 25 mg psilocybin will not take part in the open-label study phase.

If they are well enough to do so, subjects who received the full dose of psilocybin will have anxiety, depression, quality of life and spirituality measured again two months after the second experimental session. Subjects who received active placebo psilocybin will have anxiety, depression, quality of life and spirituality measured two months after the second open-label psilocybin-assisted session.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Stage IV melanoma with a life expectancy of one year or less
* Meet diagnostic criteria for anxiety on the SCID, or a score of 8 or higher on the HADS Anxiety score.
* Diagnosis must be a new diagnosis of anxiety subsequent to diagnosis with melanoma.
* Are 18 years or older
* Live with another adult who is their primary caregiver, who can also provide transportation to and from the cancer center for each experimental session and who also consents to take part in a parallel investigation of anxiety and depression in primary caregivers. The same caregiver may remain overnight with participants after each psilocybin session.
* Have a Mini-Mental State Exam score of 27 or higher, an indication of mental functioning.
* Are willing to commit to medication dosing, experimental sessions with overnight stay, traveling to follow-up sessions, and to complete the evaluation
* Are willing to refrain from taking any anti-depressants during the study period.
* Are willing to refrain from taking any benzodiazepines during the 24 hours preceding each scheduled psilocybin, placebo, or open label session.
* Are able to communicate in English.

Exclusion Criteria:

* Meet DSM-IV criteria for bipolar disorder, schizophrenia, or other psychotic disorders.
* Meet DSM-IV criteria for abuse of or dependence on any substance (other than caffeine or nicotine) in the past 60 days.
* Have first-degree relatives (as parent or full sibling) with past or present psychiatric disorders, including schizophrenia, bipolar affective disorder and other psychoses, but excluding mood disorders.
* Cannot have a current diagnosis of anxiety disorder that predates diagnosis with melanoma.
* Have used psilocybin or psilocybin-containing mushrooms within the past year.
* Require concomitant treatment with anti-psychotic medications, prescribed for the management of either psychiatric symptoms or nausea. The restriction on 5HT2C/5HT3 antagonists is applicable for 24 hours before and including the day of the study.
* Are cachectic [exhibiting signs of wasting] as indicated by loss of 10% or greater of their total weight.
* Have been diagnosed with primary or metastatic cancer of the CNS confirmed by MRI, within 6 weeks of participation in the study.
* Have uncontrolled hypertension.
* Have baseline laboratory values indicative of severely compromised hepatic function, indicated by unacceptable levels of alkaline phosphatase (ALP) above 750 U/L. Participants must also have laboratory blood screening indicating ALP below 750 U/L immediately prior to administration of psilocybin.
* Are women who are pregnant or nursing, or of child bearing potential and are not practicing an effective means of birth control.
* Are reasonably judged to present a serious suicide or homicide risk or who are likely to require psychiatric hospitalization during the course of the study.
* Are unable to fully understand the potential risks and benefits of the study and give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | Baseline, 1st non-drug intro psychotherapy, day of psilocybin-assited psychotherapy, non-drug psychotherapy between experimental sessions, day of psilocybin-assisted session 2, two weeks after second psilocybin-assisted session

SECONDARY OUTCOMES:
Spielberger-State-Trait Inventory (STAI) | Baseline, 1st intro psychotherapy, day of experimental session 1, non-drug psychotherapy between experimental sessions, day of experimental session 2, two weeks after experimental session 2
Hamilton Anxiety Rating Scale | Baseline, non-drug psychotherapy between sessions, two weeks after second experimental session
Natural killer (NK) cell count | Day after experimental session 1, day after experimental session 2
European Organization For Research and Treatment of Cancer; Quality of Life Questionnaire-C15 | Baseline, 1st intro psychotherapy, day of experimental session 1, non-drug psychotherapy between experimental sessions, day of experimental session 2, two weeks post second experimental session
Hamilton Depression Rating Scale | Baseline, non-drug psychotherapy in between experimental sessions, two weeks after second experimental session
Functional Assessment of Chronic Illness Therapy-spirituality | Baseline, first intro psychotherapy sesison, day of experimental session 1, non-drug psychotherapy between experimental sessions, day of experimental session 2, two weeks after second experimental session

CONTACTS AND LOCATIONS:
Overall Officials: Sameet Kumar, Ph.D, Principal Investigator — Psycho-oncologist, Mount Sinai Comprehensive Cancer Center
Locations (1):
- Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida, United States